CLINICAL TRIAL: NCT03761238
Title: Early Liver Support With MARS in Post-hepatectomy Liver Failure: a Randomized, Multicentre Trial
Brief Title: Early Liver Support With MARS in Post-hepatectomy Liver Failure
Acronym: ELISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stefan Gilg, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Stefan Gilg, MD, PhD, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELISH
Record Dates: First submitted 2018-11-20; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Liver Failure as A Complication of Care
Keywords: Molecular Adsorbent Recirculating System; post-hepatectomy liver failure; liver dialysis; post-hepatectomy liver dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard medical treatment + MARS (Experimental): Patients assigned to the control arm will receive standard medical treatment (SMT) and liver dialysis using Molecular Adsorbent Recirculating System (MARS).
  Interventions: Device: Molecular Adsorbent Recirculating System
- Standard medical treatment (Active Comparator): Patients assigned to the control arm will receive standard medical treatment (SMT) as specified in the study protocol.
  Interventions: Other: Standard medical treatment (SMT)

INTERVENTIONS:
Device: Molecular Adsorbent Recirculating System — MARS therapy will start within 24-48 h after randomization and be given on 3 consecutive days in sessions of 8-12 h. The patients are observed for 2 days following the last session, with focus on bilirubin INR and signs of encephalopathy, and can thereafter receive 3 additional sessions in case of no or partial response to treatment.
  Other Names: MARS 1116/1 - X-MARS
  Arms: Standard medical treatment + MARS
Other: Standard medical treatment (SMT) — Patient management and standard medical treatment (SMT) as specified in the study protocol.
  Arms: Standard medical treatment

SUMMARY:
This is a prospective, randomized, open-label, multicentre study involving European centers with experience in the management of PHLF to assess the impact of early liver support with MARS on survival in patients with post-hepatectomy liver failure (PHLF).

DETAILED DESCRIPTION:
PHLF is a major risk factor for mortality in patients who underwent major hepatectomy. A specific treatment is yet not available. In a primary proof-of-concept study, it was shown that it is safe and feasible to use MARS in patients with PHLF early after hepatectomy. Survival was superior to a historical control group.

This study will include patients with early, primary PHLF (based on the 50:50 criteria) after major liver surgery. Patients will be randomized 1:1 to receive standard treatment alone or standard treatment + liver dialysis using the Molecular Adsorbent Recirculating System (MARS). Relevant outcome along with several physiological parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected for major liver surgery (4 or more Couinaud segments) or patients undergoing a 2nd, 3rd or 4th hepatic resection. Pre-operative chemotherapy and/or biological agents are allowed.
* Primary PHLF occurring early after surgery defined by the 50:50 criteria (from PO day 5 to day 14) or by the presence of hepatic encephalopathy grade 2 or more and the 50:50 criteria (from PO day 3 to 4).
* Written informed consent.

Exclusion Criteria:

* ALPPS (Associating Liver Partition and Portal vein Ligation for Staged hepatectomy) procedure.
* In patients with chronic liver disease presence of significant portal hypertension (hepatic venous pressure gradient ≥ 10 mmHg and/or Fibroscan ≥ 21kPa) prior to surgical intervention.
* Any contraindication for MARS therapy such as uncontrolled active bleeding, platelet counts <20.000 /µl or uncontrolled infection (presence of fever or adequate antibiotic therapy for less than 48h), septic shock, haemodynamic instability requiring inotropic support (noradrenaline > 1mg/h).
* PHLF occurring after post operative day 14.
* Secondary PHLF: post-operative liver failure secondary to vascular (outflow or inflow thrombosis) or septic problems.
* Persistant biliary complications (infected biloma, main biliary tree damage).
* Inability or unwilling of the patient or family to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
60 day survival | From randomization to death from any cause, assessed up to 60 days postop
  Overall survival rate from time of randomization to death from any cause

SECONDARY OUTCOMES:
28 day survival | From randomization to death from any cause, assessed up to 28 days post-op
  Overall survival rate from time of randomization to death from any cause.
90 day survival | From randomization to death from any cause, assessed up to 90 days postop
  Overall survival rate from time of randomization to death from any cause.
6 month survival | From randomization to death from any cause, assessed up to 6 months postop
  Overall survival rate from time of randomization to death from any cause.
1 year survival | From randomization to death from any cause, assessed up to 1 year.
  Overall survival rate from time of randomization to death from any cause.
Impact of MARS therapy on liver function | From randomization up to 1 year.
  Impact of MARS therapy on liver function according to Child Pugh score (grade A, B and C)
Impact of MARS therapy on liver function | From randomization up to 1 year.
  Impact of MARS therapy on liver function according to the Model for End-stage Liver Disease (MELD) score (5 groups: < 9, 10-19, 20-29, 30-39 and >40 points, lower points indicate improvement of liver function).
Impact of MARS therapy on extra-hepatic function (APACHE-II scoring) | From randomization up to 1 year.
  Impact of MARS therapy on extra-hepatic function assessed by the Acute Physiology And Chronic Health Evaluation II (APACHE II) scoring system (range 0-71 points, lower points indicate less severe disease).
Impact of MARS therapy on extra-hepatic function (SOFA scoring) | From randomization up to 1 year.
  Impact of MARS therapy on extra-hepatic function assessed by the Sequential Organ Failure Assessment (SOFA) scoring system (0-24 points, higher points indicate more severe disease).
Impact of MARS therapy on extra-hepatic function (CLIF-SOFA scoring) | From randomization up to 1 year.
  Impact of MARS therapy on extra-hepatic function assessed by the Chronic Liver Failure-Sequential Organ Failure Assessment (CLIF-SOFA) scoring system (0-24 points, higher points indicate more severe disease).
Impact of MARS therapy on splanchnic hemodynamics assessed by direct estimation of portal blood flow. | At randomization (day 0) and on day 10.
  Impact of MARS therapy on splanchnic hemodynamics assessed by direct estimation of portal blood flow (ml/min).
Impact of MARS therapy on splanchnic hemodynamics assessed by indirect estimation of portal blood flow using ultrasonography. | At randomization (day 0) and on day 10.
  Impact of MARS therapy on splanchnic hemodynamics assessed by indirect estimation of portal blood flow using ultrasonography (ml/min).
Impact of MARS therapy on splanchnic hemodynamics assessed by portal pressure measuring. | At randomization (day 0) and on day 10.
  Impact of MARS therapy on splanchnic hemodynamics assessed by portal pressure measuring.
Impact of MARS therapy on liver regeneration assessed by volumetric liver analysis using combined Computed Tomography (CT) and Magnetic Resonance Imaging (MR). | At randomization (day 0) and on days 5, 10 and 30 .
  Impact of MARS therapy on liver regeneration assessed by volumetric liver analysis using combined Computed Tomography (CT) and Magnetic Resonance Imaging (MR).
Impact of MARS therapy on liver regeneration assessed by serum levels of phosphate. | At randomization (day 0) and on days 5 and 10.
  Impact of MARS therapy on liver regeneration assessed by serum levels of phosphate.
Impact of MARS therapy on liver regeneration assessed by serum levels of alphafetoprotein. | At randomization (day 0) and on days 5 and 10.
  Impact of MARS therapy on liver regeneration assessed by serum levels of alphafetoprotein.
Impact of MARS therapy on liver regeneration assessed by serum levels of hepatocyte growth factor. | At randomization (day 0) and on days 5 and 10.
  Impact of MARS therapy on liver regeneration assessed by serum levels of hepatocyte growth factor.
Impact of MARS therapy on liver performance status. | At randomization (day 0) and on days 5 and 10.
  Impact of MARS therapy on liver performance status estimated using indocyanine green (ICG) clearance.
Impact of MARS therapy on liver toxins (bile acids) in serum and dialysate. | At randomization (day 0) and on days 5 and 10.
  impact of MARS therapy on liver toxins (ammonia, bile acids and cytokines (IL-6 and TNF-alpha)). Determinations in serum and in the dialysate.
Impact of MARS therapy on liver toxins (ammonia) in serum and dialysate. | At randomization (day 0) and on days 5 and 10.
  impact of MARS therapy on liver toxins (ammonia). Determinations in serum and in the dialysate.
Impact of MARS therapy on liver toxins (IL-6) in serum and dialysate. | At randomization (day 0) and on days 5 and 10.
  impact of MARS therapy on liver toxins (IL-6). Determinations in serum and in the dialysate.
Impact of MARS therapy on liver toxins (TNF-alpha) in serum and dialysate. | At randomization (day 0) and on days 5 and 10.
  impact of MARS therapy on liver toxins (TNF-alpha). Determinations in serum and in the dialysate.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gilg, MD PhD, Principal Investigator — Karolinska Institutet